CLINICAL TRIAL: NCT06680414
Title: The Effects of Supportive Vaccine Communication Using Motivational Interviewing on Vaccine Knowledge, Vaccine Literacy, and Vaccine Decision Processes of Pregnant Mothers: A Waiting-List Randomized Controlled Trial
Brief Title: Impact of Supportive Vaccine Communication on Vaccine Desicion Processes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Deniz Sümeyye YORULMAZ, Asst. Prof. Dr., Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ArtvinCoruhUn
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Vaccine Hesitancy
Keywords: Vaccines; pregnant woman; experimental model; randomized controlled trial
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Random assignment. Block randomization will be used in the randomization process. Randomizer.org will be used to select block combinations with six blocks. Pregnant mothers will first be stratified according to their number of pregnancies. Eligible participants will be randomly assigned to the intervention or waitlist group using the permuted block randomization method on a 1:1 basis. The waiting list group will form the second set of the research, which is planned to be attempted two months later. The participant assignment list will be generated by a non-research statistician with a random distribution sequence. Assignment confidentiality will be ensured using opaque sealed envelopes containing sequence numbers. The data analyst/statistician will be blind to the participants' group assignments.
Who Masked: Participant
Masking Description: Single blinding(Participant blinding) will be done; participants will not be told they are in the experimental or control group. A surveyor will invite pregnant mothers to the study, which will continue until the targeted sample number (58 participants) is reached. During the participant registration, the names and contact information of the mothers will be obtained; it will be stated that they will be contacted for the training process, that the training time may be extended, and that they will be given definite training. The participant registration is completed, the supportive vaccine communication process will begin. The second researcher(D-KT) in the research team will explain to the first researcher(DS-Y) that the participants are in the experimental or control group. The pregnant mothers in the control group will be assigned to the waiting list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental (Experimental): Supportive Vaccine Communication using Motivational Interviewing will be administered to the pregnant mothers in the experimental group by the researcher. The training will take place in 3-part and 6-sessions, one week apart, and each session will last approximately 40 minutes. The training will be carried out as group training with 3-5 people. Data collection forms will be applied before and after the program.
  Interventions: Other: Supportive Vaccine Communication Using Motivational Interviewing
- control (No Intervention): No intervention will be made to the pregnant mothers in the control group during the education process of the experimental group. After the training process of the pregnant mothers in the experimental group is completed and the post-test data are collected, all the interventions and training will be given to the pregnant mothers in the control group.

INTERVENTIONS:
Other: Supportive Vaccine Communication Using Motivational Interviewing — Supportive Vaccine Communication using Motivational Interviewing will be administered to the pregnant mothers in the experimental group by the researcher. The training will take place in 3-part and 6-sessions, one week apart, and each session will last approximately 40 minutes. The training will be carried out as group training with 3-5 people. Data collection forms will be applied before and after the program.
  Arms: experimental

SUMMARY:
This research will be carried out as a randomized controlled study with a waitlist in parallel design to evaluate the effect of Supportive Vaccine Communication using Motivational Interviewing on the level of vaccination literacy, vaccine knowledge, and vaccine decision thought. Research hypothesis "H0: Supportive Vaccine Communication using Motivational Interviewing does not affect vaccine decision processes (vaccine literacy, vaccine knowledge, and vaccine decision thought). At the end of the training, it is thought that the pregnant mothers in the experimental group will be different from the control group regarding vaccine literacy, vaccine knowledge, and vaccine decision-making thoughts included in the model.

DETAILED DESCRIPTION:
In determining the sample size in the study, the smallest effect size value obtained for the Vaccine Literacy Scale result in a doctoral thesis based on another model on non-pregnant mothers in the same region was taken into consideration. In this thesis, the partial eta-squared value for Critical Vaccine Literacy was determined 0.260 (Yorulmaz, 2024). For this value, 95% power and 0.05% alpha type error margin and the total sample size required to estimate the interaction effects were determined as 48. Considering the sample losses, the sample was increased by 20% (9.6 people ~ 10 people), and a total of 58 people, 29 of which were experimental and 29 control, was determined. Pregnant mothers who apply to the obstetrics and gynecology clinic of the hospital's, which are research areas, will be evaluated according to the eligibility criteria. Then, a surveyor will obtain contact information from pregnant mothers, who met the inclusion criteria, volunteered for the study, and consented, and collect pre-test. In the study, pregnant mothers will be stratified as primiparous pregnant women (first pregnancy) and multiparous pregnant women (2 and more pregnancies). Participants will be divided into experimental and control groups using blind technique, stratification, and block randomization. The supportive vaccination communication using prepared on the motivational interview method for the pregnant mothers in the experimental group will be face-to-face training. The training will be in the form of 3-part and 6-sessions (with a 1-week interval) as group training for 3-5 people, and each session will last 40 minutes on average. After the Supportive Vaccine Communication process of the pregnant mothers in the experimental group is completed, the data collection forms will be applied again to the pregnant mothers in the experimental and control groups. After the last measurement, a 3-part, and 6-session supportive vaccine communication process will be applied to the pregnant mothers in the control group in the same way and within the same scope as the experimental group.

The primary outcome expected from the study is the change in pregnant mothers' vaccine literacy, vaccine knowledge, and vaccine decision thought.

ELIGIBILITY:
Inclusion Criteria:

* To be residing in Artvin city center
* To have applied to the gynecology and obstetrics clinic of a hospital in the city center for any reason.
* T o be in the first 28 weeks of pregnancy
* Being 18 years or older
* Turkish - speaking
* Volunteering to participate in research

Exclusion Criteria:

* 1. To reside outside of Artvin city center
* 2. To be 29 weeks or older in pregnancy
* 3. Being under 18 years old
* 4. Not know to speak Turkish
* 5. Not volunteering for research

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 58 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome expected from the study is the change in pregnant mothers' vaccine literacy. | through study completion, an average of 1 year
  Vaccine Literacy Scale: The scale evaluates the level of vaccine literacy. The Vaccine Literacy Scale was developed by Ahoran et al. (2017). The scale consists of 3 sub-dimensions and 13 items: Functional, Communicative, and Critical Health Literacy. The Functional Health Literacy subscale consists of 5 items, the Communicative Health Literacy subscale consists of 5 items, and the Critical Health Literacy subscale consists of 3 items (Ahoran et al., 2017). The Turkish evaluation of the scale was made by Yorulmaz and Kocoglu-Tanyer and, the Vaccine Literacy Scale for childhood vaccinations is a valid and reliable measurement tool for Turkish culture (Yorulmaz and Kocoglu-Tanyer, 2024).

SECONDARY OUTCOMES:
The primary outcome expected from the study is the change in pregnant mothers' vaccine knowledge. | through study completion, an average of 1 year
  Vaccine Knowledge Test: The test was developed by Yorulmaz and Kocoglu-Tanyer to assess adults' vaccine knowledge. In the Vaccine Knowledge Test, there are 28 questions answered as true, false, and do not know. Expert opinion was taken while creating the Vaccine Knowledge Test, and the content validity was evaluated. The lowest score that can be obtained from the Vaccine Knowledge Test is 0, and the highest score is 28; The increase in the total score indicates that the vaccination knowledge is high.

OTHER OUTCOMES:
The primary outcome expected from the study is the change in pregnant mothers' vaccine decision thought. | through study completion, an average of 1 year
  Vaccination Decision Thought Questionnaire: This form, which was created by researchers by reviewing the literature (Bert et al., 2020; Bisset and Paterson, 2018; Damnjanovi´c et al., 2018; Garnison et al., 2023) and taking into account the stages of the Motivational Interviewing method (Miller, 2023), includes 8 questions that evaluate pregnant women's thoughts about the safety of vaccines, the possibility of vaccinating their babies, their ability to explain the vaccine to different individuals, etc. The questions in the form are answered between 0 and 10; an increase in the answer given to each question is interpreted as an increase in the thought about the safety of vaccines, an increase in vaccine acceptance intention, an increase in self-efficacy about vaccines, and an increase in the motivation to encourage a different parent to get vaccinated.

CONTACTS AND LOCATIONS:
Locations (1):
- Deniz S. Sümeyye YORULMAZ, Merkez, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ahoran et al., 2017 — https://doi.org/10.1016/j.pec.2016.11.016
- See also: Yorulmaz and Kocoglu-Tanyer, 2024 — https://link.springer.com/article/10.1007/s10389-023-01878-5
- See also: Bisset and Paterson, 2018 — https://doi.org/10.1016/j.vaccine.2018.04.013
- See also: Damnjanovi´c et al., 2018 — https://www.frontiersin.org/journals/psychology/articles/10.3389/fpsyg.2018.00735/full